CLINICAL TRIAL: NCT04626154
Title: Validation of a Non-Invasive Device for Thoracoabdominal Asynchrony-Based Respiratory Effort Assessment in Pediatric Patients
Brief Title: Thoracoabdominal Asynchrony and Respiratory Distress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ryan Carroll, Staff physician, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2019P001411
Record Dates: First submitted 2020-10-16; First posted 2020-11-12 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: We aim to enroll pediatric patients admitted to the MGH Pediatric Intensive Care Unit (PICU): 10 patients with respiratory distress and 10 patients without respiratory distress. Readings from the TAA-monitoring device will be compared to clinical assessments made by nurses and physicians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory insufficiency or distress (Active Comparator): Patients demonstrating respiratory insufficiency or distress.
  Interventions: Diagnostic Test: Objectively monitoring thoracoabdominal asynchrony
- No respiratory insufficiency or distress. (Sham Comparator): Patients NOT demonstrating respiratory insufficiency or distress.
  Interventions: Diagnostic Test: Objectively monitoring thoracoabdominal asynchrony

INTERVENTIONS:
Diagnostic Test: Objectively monitoring thoracoabdominal asynchrony — Objectively monitoring thoracoabdominal asynchrony

SUMMARY:
The investigators hypothesize that a simple 3-point tracking device that uses motion sensors attached to the abdomen and chest of a child will provide information regarding thoracoabdominal asynchrony (TAA), a major component of respiratory distress, and ultimately help guide a clinician to initiate, escalate, de-escalate, or stop respiratory support interventions.

AIMS To determine if the TAA-monitoring device can be used to detect differences in respiratory synchrony in a manner that is clinically applicable. The investigators hope that the device will detect 1) major asynchrony events in a timely manner so as to prompt clinician intervention during future use; and 2) asynchrony events that may be less visible to the naked eye that may be precursors to more severe events.

DETAILED DESCRIPTION:
Respiratory diseases are a major global cause of morbidity and mortality in children. Of patients admitted into a pediatric intensive care unit (PICU), respiratory illnesses have been identified as the leading principal admission diagnosis in every age group, accounting for 37.9% of patients under 12 months of age and 28.5% of PICU patients across all age groups. Continuous monitoring of respiratory status is important for the guidance of respiratory support escalation and de-escalation decisions in the PICU. A clinical metric that has been suggested as a signature of breathing effort is thoracoabdominal asynchrony (TAA), the non-coincident motion of the rib cage and abdomen during breathing. A reliable, objective assessment tool for continuous monitoring of respiratory effort could allow for a more complete understanding of patients' real-time respiratory status and provide an additional indication or contraindication for the utilization of various levels of respiratory support. Limiting the use of invasive ventilatory support by early detection of respiratory distress would decrease clinical risk to patients and has the potential to decrease the cost of patient stays in the PICU. The investigators have developed a non-invasive TAA-sensing device designed for use by clinicians to indirectly quantify respiratory effort among pediatric patients (henceforth referred to as the "TAA-monitoring device"). The device utilizes motion-tracking sensors that capture data that is then processed to provide a quantitative indication of a patient's respiratory status. Given the promising yet inconclusive nature of the evidence supporting the use of TAA as an indicator of respiratory effort, clinical validation of this device is a necessary step to take to support its continued development.

ELIGIBILITY:
Inclusion Criteria:

1. patients 28-days to 17-years of age
2. who have respiratory distress and those who do not have respiratory distress

Exclusion Criteria:

Hardware, clinical care, or dermal injury that would preclude the application of TAA device

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2020-10-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Objectively determine thoracoabdominal asynchrony | Over 30 - 7200 minutes
  The investigators aim to objectively measure the frequency of asynchrony over time (minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Carroll, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No